CLINICAL TRIAL: NCT04139109
Title: The Reliability and Validity of the Turkish Version of the Survey of Activities and Fear of Falling in the Elderly
Brief Title: The Turkish Version of the Survey of Activities and Fear of Falling in the Elderly
Status: Completed | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Tansu Birinci, PT, MSc Research Assistant, Istanbul University - Cerrahpasa
Other Study IDs: 287826
Record Dates: First submitted 2019-10-22; First posted 2019-10-25 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2019-10

CONDITIONS: Fall; Old Age; Debility; Fear; Activity, Motor; Participation, Patient
Keywords: accidental falls; activity restriction; fear of falling; participation restriction; psychometrics
MeSH Terms: conditions — Frailty; Motor Activity; Patient Participation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The Survey of Activities and Fear of Falling in the Elderly (SAFE) was originally developed in English to determine the level of fear of falling and its interactions with activities of daily living. The purpose of this study was to translate and cross-culturally adapt the SAFE instrument into Turkish and investigate its psychometric properties.

DETAILED DESCRIPTION:
The Survey of Activities and Fear of Falling in the Elderly (SAFE) was originally developed in English to determine the level of fear of falling and its interactions with activities of daily living. The purpose of this study was to translate and cross-culturally adapt the SAFE instrument into Turkish and investigate its psychometric properties. One hundred eleven older adults (72 females) with a mean age of 69 years (SD=7.22; range=60-87) were included. For cross-cultural adaptation, two bi-lingual translators used the back-translation procedure. Within a 5-to-7-day period after the first assessment, the participants completed the Turkish version of SAFE (SAFE-T) to evaluate test-retest reliability. Cronbach's alpha (α) was used to assess internal consistency. The correlation with the Turkish version of the Falls Efficiency Scale-International (FES-T) was determined to check the validity.

ELIGIBILITY:
Inclusion Criteria:

1. age over 60 years old
2. ability to read and write in Turkish
3. score ≥24 on the Mini-Mental State Exam
4. >3 according to the Functional Ambulation Category (FAC)
5. no pathology in visual ability and hearing

Exclusion Criteria:

1. neurologist-diagnosed dementia or Alzheimer's disease
2. ambulatory only with a wheelchair
3. amputated lower extremity

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: One-hundred eleven older adults who were admitted to the Department of Geriatrics at Istanbul Medeniyet University Goztepe Training and Research Hospital or who volunteered to participate in this study via an online form, were evaluated between January 2018 and July 2018.
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2018-01-22 (Actual); Primary Completion 2018-04-22 (Actual); Study Completion 2018-07-22 (Actual)

PRIMARY OUTCOMES:
The Survey of Activities and Fear of Falling in the Elderly | Baseline (First assessment)
  The Survey of Activities and Fear of Falling in the Elderly (SAFE), is a reliable (α = 0.95) and valid (r = 0.91) questionnaire for evaluating activity level, fear of falling, and activity restriction. SAFE assesses 11 community-based and home-based activities. SAFE is scored as the following:
  Activity level is scored as the number of activities being done. Maximum score is 11 and higher scores indicate a higher activity level.
  The fear of falling score is computed as the average worry scores across the 11 activities (or across as many of the activities that are done, i.e., if yes to A). Each activity is scored in the range 0 to 3 by recoding the answer. The recoding is described as 0=4 (Not at all worried), 1=3 (A little worried), 2=1 (Somewhat worried) and 3=1 (Very worried). In totally, higher scores indicate a greater fear of falling.
  Activity restriction is scored by counting the number of activities which is responded "less than you used to".

SECONDARY OUTCOMES:
The Survey of Activities and Fear of Falling in the Elderly | Within a 5-to-7-day period after the first assessment (Second assessment)
  The Survey of Activities and Fear of Falling in the Elderly (SAFE), is a reliable (α = 0.95) and valid (r = 0.91) questionnaire for evaluating activity level, fear of falling, and activity restriction. SAFE assesses 11 community-based and home-based activities. SAFE is scored as the following:
  Activity level is scored as the number of activities being done. Maximum score is 11 and higher scores indicate a higher activity level.
  The fear of falling score is computed as the average worry scores across the 11 activities (or across as many of the activities that are done, i.e., if yes to A). Each activity is scored in the range 0 to 3 by recoding the answer. The recoding is described as 0=4 (Not at all worried), 1=3 (A little worried), 2=1 (Somewhat worried) and 3=1 (Very worried). In totally, higher scores indicate a greater fear of falling.
  Activity restriction is scored by counting the number of activities which is responded "less than you used to".
Falls Efficiency Scale-International | Baseline (First assessment)
  Falls Efficiency Scale-International (FES-I) is a 16-item self-administered questionnaire that was designed to assess fear of falling in community-dwelling older people. It provides information on the level of concern about falls during daily living activities. Each item is rated on a four-point scale, where 1=not at all concerned, 2=somewhat concerned, 3=fairly concerned, and 4=very concerned. The total score ranges from 16 (no concern about falling) to 64 (extreme concern about falling). The Turkish version of FES-I (FES-T), which was previously reported as a reliable (α = 0.94) and valid (r = - 0.83) instrument, was used in the present study.
History of Fall | Baseline (First assessment)
  Frequency of falls in the last six months was questioned.
Leg Pain | Baseline (First assessment)
  Presence of leg pain at rest and during activity was questioned.

CONTACTS AND LOCATIONS:
Overall Officials: Burcu Ersoz Huseyinsinoglu, PhD, Study Director — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Bakırkoy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lachman ME, Howland J, Tennstedt S, Jette A, Assmann S, Peterson EW. Fear of falling and activity restriction: the survey of activities and fear of falling in the elderly (SAFE). J Gerontol B Psychol Sci Soc Sci. 1998 Jan;53(1):P43-50. doi: 10.1093/geronb/53b.1.p43. PMID 9469171
- [Background] Allison LK, Painter JA, Emory A, Whitehurst P, Raby A. Participation restriction, not fear of falling, predicts actual balance and mobility abilities in rural community-dwelling older adults. J Geriatr Phys Ther. 2013 Jan-Mar;36(1):13-23. doi: 10.1519/JPT.0b013e3182493d20. PMID 22790588
- [Background] Yardley L, Smith H. A prospective study of the relationship between feared consequences of falling and avoidance of activity in community-living older people. Gerontologist. 2002 Feb;42(1):17-23. doi: 10.1093/geront/42.1.17. PMID 11815695
- [Background] Gazibara T, Kurtagic I, Kisic-Tepavcevic D, Nurkovic S, Kovacevic N, Gazibara T, Pekmezovic T. Falls, risk factors and fear of falling among persons older than 65 years of age. Psychogeriatrics. 2017 Jul;17(4):215-223. doi: 10.1111/psyg.12217. Epub 2017 Jan 27. PMID 28130862
- [Derived] Ersoz Huseyinsinoglu B, Tufekcioglu Z, Birinci T, Demirdag F. The Reliability and Validity of the Turkish Version of the Survey of Activities and Fear of Falling in the Elderly. J Geriatr Phys Ther. 2021 Apr-Jun 01;44(2):E132-E137. doi: 10.1519/JPT.0000000000000260. PMID 32049753